CLINICAL TRIAL: NCT07112768
Title: The Role of LH/FSH, Testosterone, Prolactin, and Ferritin in PCOS Patients in Jordan
Brief Title: LH/FSH, Testosterone, Prolactin, and Ferritin in PCOS Patients in Jordan
Acronym: PCOS patients
Status: Completed | Type: Observational
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, Assistant professor of clinical Pharmacy, Al-Ahliyya Amman University
Other Study IDs: Al-Ahliyya Amman University 1
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Five milliliters of venous blood were drawn and placed in simple test tubes for sample collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: control group (n=60), consisting control women aged 22-41 years
  Interventions: Diagnostic Test: Serum levels of LH, FSH, testosterone, prolactin, and ferritin
- PCOs group: the study group (n=80), comprising women aged 20 to 41 years who were diagnosed with PCOS based on the Rotterdam criteria (2003) as assessed by obstetric and gynecology specialist
  Interventions: Diagnostic Test: Serum levels of LH, FSH, testosterone, prolactin, and ferritin

INTERVENTIONS:
Diagnostic Test: Serum levels of LH, FSH, testosterone, prolactin, and ferritin — Measurement of both hormonal and biochemical markers in Jordanian PCOs females, including Serum levels of LH, FSH, testosterone, prolactin, and ferritin)
  Other Names: LH, FSH; testosterone; prolactin; ferritin

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is a prevalent endocrine disorder impacting women of reproductive age. Characterized by chronic anovulation, hyperandrogenism, and the presence of multiple small ovarian cysts. Despite its widespread occurrence, a comprehensive study particularly within the Jordanian population remains limited. Aim of the study: The study aimed to assess the serum levels of the Luteinizing hormone (LH), Follicle stimulating hormone (FSH), LH/FSH ratio, Testosterone, Prolactin, and Ferritin in Jordanian women diagnosed with PCOS

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is a prevalent endocrine disorder impacting women of reproductive age. Characterized by chronic anovulation, hyperandrogenism, and the presence of multiple small ovarian cysts. Despite its widespread occurrence, a comprehensive study particularly within the Jordanian population remains limited. Aim of the study: The study aimed to assess the serum levels of the Luteinizing hormone (LH), Follicle stimulating hormone (FSH), LH/FSH ratio, Testosterone, Prolactin, and Ferritin in Jordanian women diagnosed with PCOS. Materials and Methods: A total 80 women aged between 20-41 years with confirmed PCOS diagnosis and 60 age matched healthy control were enrolled. Participant completed a structured questionnaire and provided informed consent .Blood samples were collected for measurement of LH, FSH, LH/FSH ratio, testosterone, prolactin, and ferritin levels using standardized laboratory protocol. Results: There were significant differences between the PCOS and control groups in the levels of LH, FSH, LH/FSH ratio, total testosterone, prolactin, and ferritin (p<0.05 for all). Specifically, the PCOS group showed higher levels of LH, testosterone, prolactin, and ferritin, while FSH levels were significantly lower. Additionally, positive correlations were observed between LH and testosterone, FSH and prolactin, and between ferritin and both LH and the LH/FSH ratio. Conclusions: The altered hormonal and biochemical profiles observed in PCOS patients emphasize the role of these biomarkers in diagnosing and understanding the pathophysiology of PCOS. These findings could support better clinical management and inform future research, particularly in the Jordanian patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-45 PCOS diagnosed females Jordanian

Exclusion Criteria:

* younger than 20 older than 45 Non -Jordanian

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — (n=140) females were included in the current study which were subdivided into two groups: the study group (n=80), comprising women aged 20 to 41 years who were diagnosed with PCOS based on the Rotterdam criteria (2003) as assessed by obstetric and gynecology specialist [14]; and the control group (n=60), consistening control women aged 22-41
Study Population: (n=140) females were included in the current study which were subdivided into two groups: the study group (n=80), comprising women aged 20 to 41 years who were diagnosed with PCOS based on the Rotterdam criteria (2003) as assessed by obstetric and gynecology specialist ; and the control group (n=60), consistening control women aged 22-41
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Hormonal level | 3 months
  Serum levels of LH, FSH, testosterone, prolactin
Biochemical marker | 3 months
  Serum level of Ferrtin

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Ahliyya Amman University, Amman, Amman Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
The consent forms